CLINICAL TRIAL: NCT03986086
Title: A Phase 1/2 Study of MPH966, an Oral Neutrophil Elastase Inhibitor, for Prevention of Graft-versus-host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: MPH966 for Prevention of Graft-versus-host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Nelson Chao (Other)
Collaborators: Mereo BioPharma (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Nelson Chao, Donald D. and Elizabeth G. Cooke Cancer Research Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00102362
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MPH966 (Experimental): Participants receive MPH966 at RP2D tablet orally twice daily from the start of conditioning chemotherapy through 45 days post transplant.
  Interventions: Drug: MPH966
- Placebo (Placebo Comparator): Participants receive MPH placebo tablet matching MPH966 orally twice daily from the start of conditioning chemotherapy through 45 days post transplant.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MPH966 — RP2D tablet
  Other Names: alvelestat
  Arms: MPH966
Drug: Placebo — MPH966 placebo table
  Arms: Placebo

SUMMARY:
The purpose of this study is evaluate the safety and tolerability of MPH966, a neutrophil elastase inhibitor, and its ability to prevent graft-versus-host disease after hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
Phase 1 is a 3+3 dose escalation study to determine the safety and recommended phase 2 dose (RP2D) of MPH966 in patients undergoing allogeneic hematopoietic stem cell transplantation (HCT). We will evaluate up to 4 doses: 60 mg po bid, 120 mg po bid, 180 mg po bid, and 240 mg po bid. Safety, tolerability, and efficacy will be assessed in real time and pharmacokinetics and pharmacodynamics after each dose cohort before escalating to the next cohort.

Phase 2 is a randomized, double-blind, placebo-controlled study to determine the clinical efficacy of MPH966 vs. placebo in preventing acute graft-versus-host disease (GVHD) after HCT, using the RP2D as determined by the phase 1 trial.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures
2. Plan to undergo allogeneic HCT for any cancer or non-cancer illness with a planned cell dose of ≥2 x 106 CD34/kg using peripheral blood stem cells.
3. Plan to receive a myeloablative conditioning regimen (see 4.3.1).
4. Plan to receive GVHD prophylaxis with tacrolimus and methotrexate.
5. Having a donor who is a 10 of 10 HLA match;
6. Karnofsky Performance Scale KPS ≥60
7. Willing to abstain from sexual activity or use two methods of birth control while on study drug and for 5 half-lives (4 days) after last dose.

Exclusion Criteria:

1. If female, pregnant or nursing.
2. Life expectancy <6 months
3. Other malignancy or neoplastic disease (i.e. aside from the malignancy for which they are undergoing HCT) within the past 5 years with the exception of treated basal/squamous cell skin carcinoma or treated cervical cancer in situ
4. Clinically significant active infection within 1 week of starting study drug
5. Any of the following organ system function criteria:

   1. Cardiac: Ejection fraction ≤40% or myocardial infarction within 6 months of transplant or QTc >450 msec for males and >470 msec for females or other EKG abnormality which in the opinion of the investigator may put the subject at risk or interfere with study assessments
   2. Renal: Creatinine clearance (CLcr) ≤ 60 mL/min as estimated by the Cockcroft-Gault equation
   3. Pulmonary: FEV1, FVC, or corrected DLCO ≤40% predicted (forced expiratory volume in 1 second; forced vital capacity; and diffusing capacity of the lung for carbon monoxide, respectively)
   4. Hepatic: Total bilirubin >1.5 x (in the absence of known inherited hyperbilirubinemia, e.g. Gilbert's) and/or aspartate transaminase (AST)/alanine transaminase (ALT) >3 x upper limit of institutional normal for age (grade 2 or higher) and/or INR >1.5 (unless on anticoagulant), or history or evidence of cirrhosis (e.g. esophageal varices, ascites, or hepatic encephalopathy) or other chronic liver disease (e.g. Wilson's disease, autoimmune liver disease, primary biliary cirrhosis, etc.). Abnormalities in platelet number or albumin will not be considered exclusion criteria given that these are often due to the hematologic malignancy for which the patient is undergoing HCT rather than actual liver dysfunction
   5. Uncontrolled infection, including detection of hepatitis B virus (HBV) or hepatitis C virus (HCV) by serology or nucleic acid testing or HIV by polymerase chain reaction (PCR)

   i. Treated HBV/HCV/HIV with documented clearance is ok f. Other significant organ dysfunction (cardiac, pulmonary, renal, metabolic or central nervous system) that is uncontrolled and may interfere with study completion
6. Any significant medial history of alcohol abuse within 3 months of starting study drug and/or unwillingness to abstain for the duration of the study and follow up periods
7. Prior (within 30 days) or concomitant use of another neutrophil elastase inhibitor (e.g. alpha-1 antitrypsin)
8. Plan for in vivo or ex vivo T cell depletion.
9. Participated in another clinical study involving an investigational drug or device within 30 days or 5 half-lives prior to planned start of MPH966/placebo, or scheduled to participate in another clinical study involving an investigational drug or device within Day 100 of transplant

   1. If the patient develops GVHD within the first 100 days, they are allowed to enroll on trials of investigational drugs to treat GVHD provided they come off of this study.
   2. Enrollment in biorepository or supportive care trials that do not involve investigational drugs or devices is allowed
10. Any clinically relevant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis at visit, which in the opinion of the Investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study
11. Low or intermediate risk acute leukemia in first complete remission, chronic myeloid leukemia in first chronic phase, and any benign (non-malignant) disorders (phase 1 dose-escalation portion only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2-4 acute Graft vs Host Disease (GVHD) requiring systemic therapy | day 100

SECONDARY OUTCOMES:
Incidence of grade 2-4 acute GVHD | day 100
Incidence of grade 3-4 acute GVHD | day 100
Incidence of grade 2-4 acute GVHD | month 6
Incidence of grade 3-4 acute GVHD | month 6
Kaplan-Meier analysis of time-to-event: percentage of participants who develop grade 2-4 acute GVHD by visit | day 0 and 100 days, 6 months
Kaplan-Meier analysis of time-to-event: percentage of participants who develop grade 3-4 acute GVHD by visit | Day 0 and day 100, month 6
Incidence of chronic GVHD | month 6
Incidence of chronic GVHD | month 12
Kaplan-Meier analysis of time-to-event: percentage of participants who develop chronic GVHD | Day 0 and month 6, 12
  Time to event distributions estimated by the Kaplan-Meier method
Incidence of GVHD-free survival | month 6
  GVHD-free survival is defined as freedom from GVHD requiring systemic steroids
Incidence of GVHD-free survival | month 12
  GVHD-free survival is defined as freedom from GVHD requiring systemic steroids
Incidence of relapse-free survival | month 6
  Relapse-free survival is defined as freedom from relapse
Incidence of relapse-free survival | month 12
  Relapse-free survival is defined as freedom from relapse
Incidence of bacterial infections | Day 100
Incidence of fungal infections | Day 100
Incidence of viral infections | Day 100
Incidence of overall infections | Day 100
Incidence of bacterial infections | 6 months
Incidence of fungal infections | month 6
Incidence of viral infections | month 6
Incidence of overall infections | month 6
Incidence of bacterial infections | month 12
Incidence of fungal infections | month 12
Incidence of viral infections | month 12
Incidence of overall infections | month 12
Kaplan-Meier analysis of time-to-event: percentage of participants who develop bacterial infections | Day 0 and day 100, month 6,12
Kaplan-Meier analysis of time-to-event: percentage of participants who develop fungal infections | Day 0 and day 100, month 6,12
Kaplan-Meier analysis of time-to-event: percentage of participants who develop viral infections | Day 0 and day 100, month 6,12
Kaplan-Meier analysis of time-to-event: percentage of participants who develop overall infections | Day 0 and day 100, month 6,12
Incidence of relapse | month 6
Incidence of relapse | month 12
Kaplan-Meier analysis of time-to-event: percentage of participants who relapse | Day 0 and month 6,12
Incidence of non-relapse mortality | month 6
  Non-relapse mortality is defined as death while in remission from the primary disease
Incidence of non-relapse mortality | month 12
  Non-relapse mortality is defined as death while in remission from the primary disease
Kaplan-Meier analysis of time-to-event: percentage of participants who experience non-relapse mortality | Day 0 and month 6,12
  Non-relapse mortality is defined as death while in remission from the primary disease
Incidence of hospital re-admission | Day 100
Incidence of hospital re-admission | month 6
Incidence of hospital re-admission | month 12
Kaplan-Meier analysis of time-to-event: percentage of participants who are re-admitted to the hospital | Day 0 and day 100, month 6,12
Length of hospital re-admission | Day 100
Length of hospital re-admission | month 6
Length of hospital re-admission | month 12
Incidence of intensive care unit (ICU) admission | Day 100
Incidence of intensive care unit (ICU) admission | month 6
Incidence of intensive care unit (ICU) admission | month 12
Kaplan-Meier analysis of time-to-event: percentage of participants who are admitted to ICU | Day 0 and month 6,12
Length of intensive care unit (ICU) admission | Day 100
Length of intensive care unit (ICU) admission | month 6
Length of intensive care unit (ICU) admission | month 12
Length of stay in days between transplant and discharge to home | Day 0 until discharge from hospital, up to 100 days
  To determine the length of stay between transplant (Day 0) and discharge to home for those alive to be discharged home
Quality of life as measured by the FACT-BMT assessment | day 30
Quality of life as measured by the FACT-BMT assessment | day 100
Quality of life as measured by the EQ 5D-5L assessment | Day 30
Quality of life as measured by the EQ 5D-5L assessment | Day 100
Quality of life as measured by the Lorig Self-Efficacy assessment | Day 30
Quality of life as measured by the Lorig Self-Efficacy assessment | Day 100
Quality of life as measured by the PG-SGA (patient-generated subjective global assessment) | day 30
Quality of life as measured by the PG-SGA (patient-generated subjective global assessment) | day 100
Quality of life as measured by the PROMIS-Depression assessment | day 30
Quality of life as measured by the PROMIS-Depression assessment | day 100
Quality of life as measured by the PROMIS-Anxiety assessment | Day 30
Quality of life as measured by the PROMIS-Anxiety assessment | Day 100
Quality of life as measured by the PROMIS-Social Isolation assessment | Day 30
Quality of life as measured by the PROMIS-Social Isolation assessment | Day 100
Quality of life as measured by the PROMIS-Emotional Support assessment | day 30
Quality of life as measured by the PROMIS-Emotional Support assessment | Day 100
Quality of life as measured by the PROMIS-Cognitive Function assessment | Day 30
Quality of life as measured by the PROMIS-Cognitive Function assessment | Day 100
Quality of life as measured by the PROMIS-Physical Function assessment | Day 30
Quality of life as measured by the PROMIS-Physical Function assessment | Day 100
Rate of grade 2 or higher adverse events, causally related during treatment period | Day 75
Rate of grade 2 or higher adverse events, causally related during follow up period | Year 1
Rate of grade 2 or higher adverse events, non related during treatment period | Day 75
Rate of grade 2 or higher adverse events, non related during follow up period | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke University Health System (DUHS)
Locations (1):
- Duke University Adult Bone Marrow Transplant Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No